CLINICAL TRIAL: NCT05914935
Title: Safety、Tolerability、Pharmacokinetics and Initial Efficacy of Recombinant L-IFN Adenovirus Injection in the Treatment of Recurrent Glioblastoma：an Open-label, Single-arm, Single-center, Multi-dose Investigator-initiated Clinical Trial
Brief Title: Safety and Tolerability Study of Recombinant L-IFN Adenovirus Injection in Patients With Recurrent Glioblastoma
Acronym: YSCH-01
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Binhai Hospital of Fujian Medical University (Other)
Collaborators: Shanghai Yuansong Biotechnology Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YSCH-01-001
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Recurring Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant L-IFN adenovirus injection and Ommaya reservoir (Experimental): Recombinant L-IFN adenovirus injection was locally injected through the Ommaya reservoir.A single injection dose of 5.0×10^10 VP (total dose per injection) was administered during the treatment period.
  Interventions: Drug: Recombinant L-IFN adenovirus injection

INTERVENTIONS:
Drug: Recombinant L-IFN adenovirus injection — The Ommaya reservoir was surgically implanted, and multiple intracapsular injections were given medicine. On the second day after Ommaya reservoir implantation, CT examination confirmed that the implantation was successful, and the experimental drug injection was started.
  Other Names: YSCH-01; Oncolytic adenovirus

SUMMARY:
The target subjects were patients with histologically or cytologically confirmed recurrent glioblastoma.Six subjects were expected to be enrolled,the number of subjects will be adjusted according to the course and outcome of the trial.The aim of this study was to evaluate the safety and tolerability of recombinant L-IFN adenovirus injection in the treatment of patients with recurrent glioblastoma, and to determine the registered clinical recommended dose and dosing regimen.

DETAILED DESCRIPTION:
The IIT clinical study of recombinant L-IFN adenovirus injection is planned to adopt an open-label, non-randomized, dose exploratory study design. The trial was divided into screening, treatment and maintenance periods.The Ommaya reservoir was surgically implanted, and multiple intracapsular injections were administered.The overall survival (OS), progression-free survival (PFS) and disease control rate (DCR) were used to evaluate the efficacy of recombinant adenovirus L-IFN injection in the treatment of recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1.Voluntarily sign the informed consent and follow the requirements of the protocol; 2.18 years old ≤ age ≤75 years old, male or female; 3. Expected survival time ≥12 weeks; 4.KPS score ≥50 before treatment; 5. Patients with pathologically and/or cytologically confirmed glioblastoma; After conventional radiation and/or systemic therapy, the disease recurred. PETCT/MRI of the head within 14 days before screening confirmed at least one enhancement lesion ≥1 cm in length.

6. The patient has recovered from the toxic effects of the last treatment before the first dose (CTCAE≤1, except for special conditions such as "alopecia" and "pigmentation"), and the corresponding AE is judged by the investigator to be not a safety risk; 7. Organ and bone marrow function levels must meet the following requirements:

1. Bone marrow: Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90 g/L, and no platelet or red blood cell transfusion within 14 days before the first dose; No blood transfusion or biological response regulators (such as granulocyte stimulating growth factor, erythrocyte growth factor, interleukin-11, etc.) within 14 days before the first dose;
2. Liver function: No history of cirrhosis (Child-Pugh class B, C decompensated cirrhosis) Patients without liver metastasis were required to have serum total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN. Patients with liver metastasis required TBIL ≤1.5×ULN, ALT and AST≤5×ULN;
3. Renal function: serum creatinine ≤1.5×ULN or creatinine clearance ≥50 ml/ minute (Cockcorft-Gault formula) Qualitative urine protein ≤1+; If urinary protein qualitative ≥2+，24-hour urinary protein quantitative test is required. The investigators determined the enrollment according to the examination results.
4. Coagulation: prothrombin time (PT) ≤1.5 times ULN An international normalized ratio (INR) of 1.5×ULN or less and an activated partial thromboplastin time (APTT) of 1.5×ULN or less (except for those receiving therapeutic anticoagulants); 8. Female participants of childbearing age must have taken a serum pregnancy test with a negative result within 3 days before starting study medication and be willing to use a medically approved, highly effective contraceptive (e.g., IUD, contraceptive pill, or condom) during the study and for 5 months after last administration of study medication; For male subjects whose partner was a woman of childbearing age, consent was given to use an effective method of contraception for the duration of the study and for 5 months after the last study dose.

Exclusion Criteria:

1. Previous or current history of other types of malignant tumors, except for the following:

   1. radical cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma, or cervical cancer in situ;
   2. second primary cancer that has been cured with no recurrence within 5 years;
2. Known allergy to the study drug or any of its excipients, or a history of unexplained severe allergic reaction;
3. Any contraindications to gadolinium contrast-enhanced MRI, such as personal use of a pacemaker, infusion pump, or allergy to MRI contrast media;
4. Any contraindications to implantation of Ommaya reservoir;
5. Received any of the following treatments or medications before the first study treatment:

   1. major surgery or major trauma within 4 weeks before the first study drug. (Major surgery is defined as any invasive procedure that involves extensive resection or that requires opening of mesothelial cell barriers (e.g., pleural space, peritoneum, meninges). However, biopsies needed for diagnosis were permitted. Severe trauma is a wound, ulcer or fracture that does not heal;
   2. administration of live attenuated vaccine within 4 weeks before or planned for the duration of the first study drug;
   3. medium (adult) drug treatment with anti-tumor indications within 2 weeks before the first study drug treatment;
   4. antineoplastic therapy (including chemotherapy, radiotherapy, immunotherapy, targeted therapy, biological therapy or tumor embolization) within 4 weeks before the first dose; For oral fluorouracil and endocrine therapy, drug withdrawal ≤2 weeks; In the case of nitrosourea, mitomycin or monoclonal antibody, drug withdrawal ≤6 weeks. If washout time is insufficient due to schedule or PK characteristics of the drug, it needs to be discussed with the partner;
6. Patients with symptoms, disseminated to viscera, and risk of life-threatening complications in a short period of time, patients with pleural effusion, peritoneal effusion, and pericardial effusion who underwent puncture and drainage within three weeks before the first administration;
7. Subjects with active or preexisting autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.) or those at high risk (e.g., organ transplant recipients requiring immunosuppressive therapy). However, subjects with the following conditions were allowed:

   1. patients with type I diabetes who are stable on fixed doses of insulin;
   2. autoimmune hypothyroidism with hormone replacement therapy only;
   3. skin conditions requiring no systemic treatment (e.g. eczema, rashes covering less than 10% of the body surface, psoriasis without eye symptoms, etc.);
   4. patients who have resolved childhood asthma/allergy without intervention in adulthood;
8. Cardiovascular disease within 6 months before screening meets any of the following criteria:

   1. congestive heart failure with New York Heart Association (NYHA) class Ⅱ or above; Left ventricular ejection fraction (LVEF) < 50%;
   2. severe arrhythmias requiring medical treatment;
   3. QTcF (Fridericia's formula) > 450 msec in a man or > 470 msec in a woman, or the presence of risk factors for torsdes pointes, such as hypokalemia, a family history of long QT syndrome, or a family history of arrhythmias (e.g., the Wolff-White syndrome), as judged by the investigator to be clinically significant;
   4. a history of myocardial infarction or severe/unstable angina within 6 months before treatment;
   5. a history of thromboembolic events of grade ≥3 within the past 2 years or receiving thrombolytic or anticoagulant therapy due to a high risk of thrombosis;
9. Patients with sudden lung disease, interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, etc. which could not be controlled after treatment, except for local interstitial pneumonia induced by radiotherapy;
10. Uncontrolled systemic diseases, such as diabetes (fasting blood glucose ≥13.3mM), hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), etc.;
11. Have a history of human immunodeficiency virus infection or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or stem cell transplantation; Except for those who do not require immunosuppressive therapy, such as corneal transplantation;
12. Evidence of active infection:

    1. Hepatitis B (HBsAg positive, HBV-DNA≥500IU/ml and abnormal liver function);
    2. Hepatitis C (HCV-Ab positive, HCV-RNA higher than the detection limit of analytical method and abnormal liver function);
    3. Systemic use of anti-infective agents for ≥7 days within 4 weeks before the first dose or unexplained fever > 38.5°C during screening/before the first dose (according to the investigator's judgment, fever caused by cancer could be enrolled);
    4. Patients with active pulmonary tuberculosis infection detected by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year before enrollment but without regular treatment;
13. A definite history of a previous neurological or mental disorder or a known history of psychotropic substance abuse, alcohol abuse or drug use;
14. Received any investigational drug within 4 weeks before the first dose or was enrolled in another clinical study (except if the patient was enrolled in an observational, noninterventional clinical study or was in the follow-up period of an interventional clinical study; or more than 5 half-lives of the last study medication);
15. Women who are pregnant or lactating, or who have a positive baseline pregnancy test;
16. Patients deemed by the investigator to be ineligible for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Up to 28 days
  To define the maximum tolerated dose (MTD) of intratumoral administration of Recombinant L-IFN adenovirus injection in humans with malignant tumors
Safety and tolerability assessed by Adverse Events (AEs) | Up to 6 months
  An AE is any untoward medical occurrence in a subject administered an investigational product (IP), and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP

SECONDARY OUTCOMES:
Overall survival (OS) | 3.5 years
  Months alive following treatment as measured during periodic study visits
Presence of neutralizing antibodies of antidrug antibodies (ADAs) development | Up to 6 months
  To evaluate the immunogenicity of Recombinant L-IFN adenovirus injection given as single agent post injection
Quality of life (QOL) | 18 months
  To measure quality of life (QOL) baseline assessment and any changes over time，EORTC QLQ-C30 scale was used for assessment，except for items 29 and 30, all items in QLQ-C30 scale are reverse items (the higher the value, the worse the quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Dezhi Kang, PhD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Binhai Hospital of Fujian Medical University, Fujian, Fujian, China